CLINICAL TRIAL: NCT01434290
Title: A Randomized Phase II Trial of Hypofractionated Radiotherapy for Favorable Risk Prostate Cancer
Brief Title: Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0938; CDR0000703580; NCI-2011-03629 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Radiation Toxicity; Sexual Dysfunction
Keywords: radiation toxicity; sexual dysfunction; psychosocial effects of cancer and its treatment; adenocarcinoma of the prostate; stage I prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 Fractions (Experimental): 36.25 Gy IMRT in 5 fractions over two and a half weeks
  Interventions: Radiation: 36.25 Gy IMRT
- 12 Fractions (Experimental): 51.6 Gy IMRT in 12 fractions over two and a half weeks
  Interventions: Radiation: 51.6 Gy IMRT

INTERVENTIONS:
Radiation: 36.25 Gy IMRT — 36.25 Gy in 5 fractions of 7.5 Gy twice a week over 15-17 days. A minimum of 72 hours and a maximum of 96 hours will separate each treatment. IMRT or similar techniques that use inverse treatment planning or protons are required.
  Arms: 5 Fractions
Radiation: 51.6 Gy IMRT — 51.6 Gy in 12 fractions of 4.3 Gy 5 days a week over 16-18 days. IMRT or similar techniques that use inverse treatment planning or protons are required.
  Arms: 12 Fractions

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Given radiation therapy in different ways may kill more tumor cells.

PURPOSE: This randomized phase II trial studies radiation therapy to see how well it works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate that 1-year health-related quality of life (HRQOL) for at least one hypofractionated arm is not significantly lower than baseline as measured by the Bowel and Urinary domains of the Expanded Prostate Cancer Index Composite (EPIC) instrument.

Secondary

* To estimate the degree of change in HRQOL in each arm for the Sexual and Hormonal EPIC domains and the Utilization of Sexual Medications/Devices from baseline to 1 year, 2 years, and 5 years.
* To estimate the degree of change in global HRQOL in each arm as measured by the Euro Quality of Life, 5 dimensions (EQ-5D) from baseline to 1 year, 2 years, and 5 years.
* To estimate the rate of acute and late gastrointestinal (GI) and genitourinary (GU) toxicity for each arm at 1, 2, and 5 years.
* To estimate prostate-specific antigen (PSA) failure in each arm at 1, 2, and 5 years.
* To estimate disease-free survival (DFS) in each arm at 1, 2, and 5 years.
* To estimate Quality Adjusted Life Years for each arm at 1, 2, and 5 years using the EQ-5D and DFS.
* To identify genetic markers associated with normal tissue toxicities resulting from radiotherapy.
* To collect tumor tissue for biomarker studies.
* To estimate EPIC bowel and urinary HRQOL as continuous variables.

OUTLINE: This is a multicenter study. Patients are stratified according to treatment techniques/machine (all linear accelerator-based treatment [excluding cyberknife] vs cyberknife vs protons). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo hypofractionated radiotherapy using intensity-modulated radiation therapy (IMRT), cyberknife, or protons twice a week for approximately 2½ weeks (36.25 Gy total).
* Arm II: Patients undergo hypofractionated radiotherapy using IMRT, cyberknife, or protons once a day, 5 days a week, for approximately 2½ weeks (51.6 Gy total).

Patients may undergo blood and tumor tissue collection for correlative studies.

Patients may also complete the Utilization of Sexual Medications/Devices, the European Questionnaire-5D, and the Bowel and Urinary domains of the Expanded Prostate Cancer Index Composite (EPIC) questionnaires at baseline and at 1, 2, and 5 years after completion of radiation therapy.

After completion of study therapy, patients are followed-up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days of randomization

  * History/physical examination with digital rectal examination of the prostate within 60 days prior to registration
  * Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason scores 2-6 within 180 days of randomization
  * Clinical stage T1-2a (AJCC 7th edition) within 90 days of randomization
  * Prostate-specific antigen (PSA) < 10 ng/mL within 60 days prior to registration;

    * PSA should not be obtained within 10 days after prostate biopsy
* No evidence of distant metastases
* No regional lymph node involvement

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire
* No prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease-free for a minimum of 5 years (for example, carcinoma of the oral cavity is permissible; however, patients with prior history of bladder cancer are not allowed)
* No severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects

    * Laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current Center for Disease Control (CDC) definition

    * HIV testing is not required for entry into this protocol
    * Protocol-specific requirements may also exclude immuno-compromised patients

PRIOR CONCURRENT THERAPY:

* No prior radical surgery (prostatectomy), cryosurgery, or high-intensity focused ultrasonography (HIFU) for prostate cancer
* No prior pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* No prior hormonal therapy, such as luteinizing hormone-releasing hormone (LHRH) agonists (e.g., goserelin, leuprolide) or LHRH antagonists (e.g., degarelix), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g., diethylstilbestrol (DES)), or surgical castration (orchiectomy)
* No finasteride within 30 days prior to registration

  * Prostate-specific antigen (PSA) should not be obtained prior to 30 days after stopping finasteride
* No dutasteride within 90 days prior to registration

  * PSA should not be obtained prior to 90 days after stopping dutasteride
* No prior or concurrent cytotoxic chemotherapy for prostate cancer
* Patients on Coumadin or other blood-thinning agents are eligible for this study
* No concurrent 3D-conformal radiation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himu R. Lukka, MD, Principal Investigator — Margaret and Charles Juravinski Cancer Centre
Locations (37):
- United States (32):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Kaiser Permanente - Division of Research - Oakland, Oakland, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Urology Center of Colorado, Denver, Colorado
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Rothman Specialty Hospital, Bensalem, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Academic Urology Prostate Center, King of Prussia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (5):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Fractions: 36.25 Gy IMRT (intensity modulated radiation therapy) in 5 fractions over two and a half weeks
Period: Overall Study
Arm/Group | 5 Fractions | 12 Fractions
Started | 127 | 128
Completed | 119 (Eligible subjects included in analysis) | 121 (Eligible subjects included in analysis)
Not Completed | 8 | 7
Not completed — Protocol Violation | 6 | 3
Not completed — No protocol treatment | 2 | 4

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 Fractions | 12 Fractions | Total
Number analyzed (Participants) | 119 | 121 | 240
Age, Continuous [Median (Full Range); unit: years] | 64 [48 to 77] | 66 [50 to 79] | 65 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 119 | 121 | 240

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Reduction From Baseline to the One-year EPIC Bowel Domain Score That Exceeds 5 Points
Description: The co-primary endpoint is the percentage of patients with a reduction in the Expanded Prostate Cancer Index Composite (EPIC) bowel domain score from baseline to 1 year that exceeds 5 points (baseline - one year > 5). The EPIC is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal). Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. Arms are not compared to each other.
Time Frame: Baseline and one year from the end of protocol treatment
Population: Eligible patients who started protocol treatment and completed the bowel domain of the EPIC at baseline and one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 93 | 100
percentage of participants | 30.1 [20.8 to 39.4] | 28.0 [19.2 to 36.8]
Statistical Analysis 1: Comparison: 5 Fractions; ≤35% was considered acceptable, ≥55% unacceptable. Each arm analyzed separately. Average score and standard error of each arm calculated and one-sample z-test for proportion with significance level of 0.025 was used. For a given arm, if the null hypothesis of p ≤ 0.35 is rejected, then conclude that the regimen given on that arm is unacceptable. However if it not rejected for both bowel & urinary domains, then that regimen will be considered acceptable for further use in a Phase III study; Test type: Superiority; p = 0.19, One sample z-test; One-sided 0.025 significance level
Statistical Analysis 2: Comparison: 12 Fractions; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.08, One sample z-test; one-sided 0.025 significance level

2. Primary Outcome: The Percentage of Patients With Reduction From Baseline to One-year EPIC Urinary Domain Score That Exceeds 2 Points
Description: The co-primary endpoint is the proportion of patients with a reduction in the Expanded Prostate Cancer Index Composite (EPIC) urinary domain score from baseline to 1 year that exceeds 2 points (baseline - one year > 2). The EPIC is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal). Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. Arms are not compared to each other.
Time Frame: Baseline and one year from the end of protocol treatment
Population: Eligible patients who started protocol treatment and completed the urinary domain of the EPIC at baseline and one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 93 | 100
percentage of participants | 45.2 [35.4 to 55.0] | 42.0 [32.3 to 51.7]
Statistical Analysis 1: Comparison: 5 Fractions; ≤40% was considered acceptable, ≥60% unacceptable. Each arm analyzed separately. Average score and standard error of each arm calculated and one-sample z-test for proportion with significance level of 0.025 was used. For a given arm, if the null hypothesis of p ≤ 0.40 is rejected, then conclude that the regimen given on that arm is unacceptable. However if it not rejected for both bowel & urinary domains, then that regimen will be considered acceptable for further use in a Phase III study; Test type: Superiority; p = 0.18, One sample z-test; One-sided 0.025 significance level
Statistical Analysis 2: Comparison: 12 Fractions; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.38, One sample z-test; One-sided 0.025 significance level

3. Secondary Outcome: Acute and Late Gastrointestinal (GI) and Genitourinary (GU) Toxicity for Each Arm
Description: Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the adverse event (AE). The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. An acute adverse event is defined as the first occurrence of worst severity of the adverse event ≤30 days after the completion of radiation therapy (RT). The high dose RT arm of Radiation Therapy Oncology Group (RTOG) study RTOG-0126 (NCT00033631) reported 1% of patients experienced grade 3+ GI/GU acute toxicity with no patient experiencing a grade 4 or 5 toxicity. If the lower confidence interval is >1%, then that arm will be further investigated for acceptability. A late adverse event is defined as the first occurrence of worst severity of adverse event >30 days after RT completion. Arms are not compared to each other.
Time Frame: Start of protocol treatment to one year from the end of protocol treatment
Population: Eligible patients who started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 119 | 121
percentage of participants
  Acute | 1.7 [0.2 to 5.9] | 1.7 [0.2 to 5.9]
  Late | 0.8 [0.1 to 4.2] | 0.8 [0.1 to 4.2]

4. Secondary Outcome: Rate of PSA Failure
Description: Failure occurs when the PSA is first noted to be 2 ng/mL or more than the current nadir value (PSA > current nadir + 2) post RT completion. Time to PSA failure is defined as time from registration to the date of PSA failure, last known follow-up (censored), or death without PSA failure (competing risk). Rate of PSA failure is estimated by the cumulative incidence method. The protocol specified that one-, two-, and five-year rates would be reported. Arms are not compared to each other.
Time Frame: Registration to five years
Population: Eligible patients who started protocol treatment and were at risk at the given time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 119 | 121
percentage of participants
  One year | 0.0 [NA to NA] — Insufficient number of participants with events | 0.8 [0.1 to 4.1]
  Two years: number analyzed (Participants) | 118 | 115
  Two years | 0.0 [NA to NA] — Insufficient number of participants with events | 0.8 [0.1 to 4.1]
  Five years: number analyzed (Participants) | 93 | 97
  Five years | 3.4 [1.1 to 8.0] | 3.5 [1.1 to 8.0]

5. Secondary Outcome: Rate of Disease-free Survival (DFS)
Description: Disease-free survival duration is time from the date of randomization to the date of documentation of disease progression or until the date of death from any cause (censored). DFS is estimated by the Kaplan-Meier method. The protocol specified that one-, two-, and five-year rates would be reported. Arms are not compared to each other.
Time Frame: Registration to 5 years
Population: Eligible patients who started protocol treatment and were at risk at the given time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 119 | 121
percentage of participants
  One year: number analyzed (Participants) | 118 | 120
  One year | 99.2 [97.5 to 100.0] | 99.2 [97.6 to 100.0]
  Two years: number analyzed (Participants) | 118 | 115
  Two years | 99.2 [97.5 to 100.0] | 97.5 [94.7 to 100.0]
  Five years: number analyzed (Participants) | 92 | 97
  Five years | 89.6 [84.0 to 95.2] | 92.3 [87.4 to 97.1]

6. Secondary Outcome: Mean Quality Adjusted Life Years at 5 Years
Description: Quality-adjusted survival time combines disease-free survival time and quality of life as measured by the EuroQol 5-dimensional (EQ-5D) index score. It is calculated for each patient as the weighted sum of different time episodes and added up to total quality-adjusted life years . The EQ-5D measures health-related quality of life and consists of two parts, a general health visual analog scale and 5 general health questions. The latter questions are transformed into a single index score ranging from 0 (worst health state) to 1 (best health state). Arms are not compared to each other.
Time Frame: Registration to 5 years from the end of protocol treatment
Population: Eligible patients who started protocol treatment with baseline EQ-5D and at least 1 follow-up assessment (EQ-5D Index Score)
Measure: Mean (Standard Deviation); unit: quality-adjusted life years
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 90 | 85
quality-adjusted life years | 6.13 (10.55) | 4.87 (1.14)

7. Secondary Outcome: Change From Baseline in EPIC Bowel and Urinary HRQOL as Continuous Variables at One Year
Description: The EPIC is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal). Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life and a positive change from baseline indicating improvement over time. For this endpoint, in each domain, the actual change score calculated as timepoint score - baseline score will be used as the statistic.
Time Frame: Baseline and one year from the end of protocol treatment
Population: Eligible patients who started protocol treatment and completed the respective domain of the EPIC at baseline and one year
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 93 | 100
units on a scale
  1-year Bowel | 1.79 [-26.79 to 53.57] | 0 [-26.79 to 46.42]
  1-year Urinary | 0 [-25.75 to 69.42] | 0 [-47.92 to 63.91]
Statistical Analysis 1: Comparison: 5 Fractions; [Bowel one-year results] Originally the t-test was planned to test if the change in each arm is different from 0. Wilcoxon Mann-Whitney was used instead due to the normality of the data; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017
Statistical Analysis 2: Comparison: 12 Fractions; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017
Statistical Analysis 3: Comparison: 5 Fractions; [Urinary one-year results] Originally the t-test was planned to test if the change in each arm is different from 0. Wilcoxon Mann-Whitney was used instead due to the normality of the data; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017
Statistical Analysis 4: Comparison: 12 Fractions; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney); Two-side significance level of 0.017

8. Secondary Outcome: The Percentage of Patients With Reduction From Baseline at One Year in EPIC Sexual Domain Score That Exceeds 11 Points
Description: The percentage of patients with a reduction in the EPIC sexual domain score from baseline that exceeds 11 points (baseline - one year > 11). The EPIC is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal). Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. Arms are not compared to each other.
Time Frame: Baseline one year from the end of protocol treatment
Population: Eligible patients who started study treatment and completed the specified domain of the EPIC at baseline and one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 88 | 92
percentage of participants | 32.9 [23.1 to 42.7] | 30.4 [21.0 to 39.8]
Statistical Analysis 1: Comparison: 5 Fractions; ≤35% was considered acceptable, ≥55% unacceptable. Each arm analyzed separately. Average score and standard error of each arm calculated and one-sample z-test for proportion with significance level of 0.025 was used; Test type: Superiority; p = 0.39, One-sample z-test; One-sided 0.025 significance level
Statistical Analysis 2: Comparison: 12 Fractions; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.21, One sample z-test; One-side significance level of 0.025

9. Secondary Outcome: The Percentage of Patients With Reduction From Baseline at One Year in EPIC Hormonal Domain Score That Exceeds 3 Points
Description: The percentage of patients with a reduction in the EPIC hormonal domain score from baseline that exceeds 3 points (baseline - one year > 3). The EPIC is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal). Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. Arms are not compared to each other.
Time Frame: Baseline and one year from the end of protocol treatment
Population: Eligible patients who started study treatment and completed the specified domain of the EPIC at baseline and one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 90 | 97
percentage of participants | 36.7 [26.7 to 46.7] | 38.1 [28.4 to 47.8]
Statistical Analysis 1: Comparison: 5 Fractions; ≤38% was considered acceptable, ≥58% unacceptable. Each arm analyzed separately. Average score and standard error of each arm calculated and one-sample z-test for proportion with significance level of 0.025 was used; Test type: Superiority; p = 0.44, one sampe z-test; One-sided significance level of 0.025
Statistical Analysis 2: Comparison: 12 Fractions; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.53, One sample z-test; One-sided significance level of 0.025

10. Secondary Outcome: Change From Baseline in EQ-5D Scores
Description: The EQ-5D is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). Health states are defined by the combination of the leveled responses to the 5 dimensions, generating 243 health states to which unconsciousness and death are added. The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm 10-point interval scale. Worst imaginable health state is scored as 0 at the bottom of the scale, and best imaginable health state is scored as 100 at the top. The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). Change from baseline is calculated as score at the timepoint of interested - baseline score. One, 2, and 5 years will be entered when they are available. Arms are not compared.
Time Frame: Baseline and one year from the end of protocol treatment
Population: All eligible patients who started study treatment and completed the EQ-5D at baseline and the specified timepoint
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 66 | 67
units on a scale
  1-year Index Score | 0 [-0.554 to 0.200] | 0 [-0.447 to 0.603]
  1-year VAS: number analyzed (Participants) | 65 | 63
  1-year VAS | 0 [-30 to 74] | 0 [-60 to 89]
Statistical Analysis 1: Comparison: 5 Fractions; [One-year Index Score] Originally the t-test was planned to test if the change in each arm is different from 0. Wilcoxon Mann-Whitney was used instead due to the non-normality of the data. Each arm analyzed separately; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017
Statistical Analysis 2: Comparison: 12 Fractions; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017
Statistical Analysis 3: Comparison: 5 Fractions; [One-year VAS Score] Originally the t-test was planned to test if the change in each arm is different from 0. Wilcoxon Mann-Whitney was used instead due to the non-normality of the data. Each arm analyzed separately; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017
Statistical Analysis 4: Comparison: 12 Fractions; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney); Two-sided significance level of 0.017

11. Secondary Outcome: Utilization of Sexual Medications/Devices Questionnaire Response Frequences
Description: The Utilization of Sexual Medications/Devices questionaire is designed to assess the use of erectile aids among patients treated for prostate cancer. This instrument is used to complement the sexual symptom domain in the EPIC. The number of subjects responding "Yes" to the following questions are reported: "Do you have a penile prosthesis", "Have you used an medications or devices to aid or improve erections?". Arms are not compared to each other. One, 2, and 5 years will be entered when they are available.
Time Frame: Baseline and one year from the end of protocol treatment
Population: Eligible patients who started study treatment and completed the questionnaire at baseline and the specified timepoint
Measure: Number; unit: participants
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 94 | 96
participants
  Baseline penile prosthesis question | 6 | 7
  Baseline medications/devices question: number analyzed (Participants) | 91 | 94
  Baseline medications/devices question | 30 | 29
  1-year penile prosthesis question: number analyzed (Participants) | 81 | 82
  1-year penile prosthesis question | 2 | 5
  1-year Baseline medications/devices question: number analyzed (Participants) | 79 | 78
  1-year Baseline medications/devices question | 25 | 29

12. Secondary Outcome: Genetic Markers Associated With Normal Tissue Toxicities Resulting From Radiotherapy
Time Frame: Study entry to 5 years from the end of protocol treatment
Population: The biomarker data will not be obtained due to lack of funding therefore no patients have outcome measure data.
Arm/Group | 5 Fractions | 12 Fractions
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event. Eligible patients with adverse event data are included.
Arm/Group | 5 Fractions | 12 Fractions
Serious Adverse Events (participants affected / at risk) | 1/119 | 0/121
Other Adverse Events (participants affected / at risk) | 101/119 | 106/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 Fractions (N=119) | 12 Fractions (N=121)
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 Fractions (N=119) | 12 Fractions (N=121)
Constipation (Gastrointestinal disorders) | 10 | 5
Diarrhea (Gastrointestinal disorders) | 28 | 31
Fecal incontinence (Gastrointestinal disorders) | 8 | 6
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 15 | 15
Hemorrhoids (Gastrointestinal disorders) | 9 | 8
Proctitis (Gastrointestinal disorders) | 18 | 21
Rectal hemorrhage (Gastrointestinal disorders) | 13 | 5
Rectal pain (Gastrointestinal disorders) | 6 | 2
Fatigue (General disorders) | 30 | 34
Libido decreased (Psychiatric disorders) | 10 | 6
Cystitis noninfective (Renal and urinary disorders) | 17 | 20
Hematuria (Renal and urinary disorders) | 9 | 11
Renal and urinary disorders - Other (Renal and urinary disorders) | 33 | 35
Urinary frequency (Renal and urinary disorders) | 66 | 70
Urinary incontinence (Renal and urinary disorders) | 16 | 22
Urinary retention (Renal and urinary disorders) | 22 | 26
Urinary tract obstruction (Renal and urinary disorders) | 10 | 6
Urinary tract pain (Renal and urinary disorders) | 13 | 21
Urinary urgency (Renal and urinary disorders) | 39 | 47
Ejaculation disorder (Reproductive system and breast disorders) | 11 | 12
Erectile dysfunction (Reproductive system and breast disorders) | 51 | 44
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.